CLINICAL TRIAL: NCT05116436
Title: Genetic Study of Idiopathic Scoliosis in a Cohort of Families
Brief Title: Genetic Study of Idiopathic Scoliosis in a Cohort of Families (SCOGEN)
Acronym: SCOGEN
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ramsay Générale de Santé (Other)
Collaborators: European Clinical Trial Experts Network (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-A03136-51
Record Dates: First submitted 2021-11-04; First posted 2021-11-11 (Actual); Last update posted 2021-11-11 (Actual); Status verified 2021-11

CONDITIONS: Scoliosis Idiopathic
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patient with idiopathic scoliosis
  Interventions: Procedure: Blood sample; Procedure: Spine X-ray
- Healthy related patients
  Interventions: Procedure: Blood sample; Procedure: Spine X-ray

INTERVENTIONS:
Procedure: Blood sample — It will test the presence or absence of genetic mutations found in other cohorts in previous studies.
Procedure: Spine X-ray — To determine the scoliosis

SUMMARY:
This study will focus on a large cohort of multiplex families, to precisely identify candidate genes. The fact of have a large database (fifty families, collected by the principal investigator for more than two decades), will contribute to the discovery of genes of interest. It will also allow testing for the presence or absence of mutations found in other cohorts in previous studies. The main objective of this study is to identify genetic abnormalities associated with the presence and severity of idiopathic scoliosis, in families of scoliosis.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for "sick" patients:

* Presence of idiopathic scoliosis, diagnosed by a clinical examination by an orthopedic doctor and confirmed by the presence of a Cobb angle greater than 10 ° on radiographs of the spine
* Signed informed consent
* Affiliation to a social security scheme or beneficiary of such a scheme

Inclusion criteria for "healthy relatives":

* Be related to the first or second degree with at least 2 individuals suffering from idiopathic scoliosis, and whose family tree over 3 generations finds at least 3 cases of idiopathic scoliosis
* Do not present with scoliosis (clinical examination by an orthopedic doctor and x-rays of the spine).
* Affiliation to a social security scheme or beneficiary of such a scheme

Exclusion Criteria:

Non-inclusion criteria for "sick" patients:

* Be part of one of the following categories of vulnerable people: protected adults, adults unable to express their consent and not subject to a protection measure, pregnant women, parturients and nursing mothers, people deprived of their liberty, people hospitalized without consent, people admitted to a health or social establishment for purposes other than research
* Suspicion of scoliosis secondary to clinical examination

Non-inclusion criteria for "healthy relatives":

* Be part of one of the following categories of vulnerable people: protected adults, adults unable to express their consent and not subject to a protection measure, pregnant women, parturients and nursing mothers, people deprived of their liberty, people hospitalized without consent, people admitted to a health or social establishment for purposes other than research
* Discovery of scoliosis during research (if scoliosis of an idiopathic nature: patient included in the cohort of patients, if secondary scoliosis: exclusion from the family).

All patients :

Pregnancy in progress or desired with discontinuation of contraception (contraindication to the realization of x-rays).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Families : patients with idiopathic scoliosis and their relatives
Sampling Method: Non-Probability Sample
Enrollment: 43 (Estimated)
Dates: Start 2020-06-06 (Actual); Primary Completion 2021-06-06 (Actual); Study Completion 2022-06-06 (Estimated)

PRIMARY OUTCOMES:
Presence of a mutated allele in scoliosis patients versus their healthy relatives. | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Clinique Maussins-Nollet, Paris, France